CLINICAL TRIAL: NCT07074795
Title: Nitrous Oxide During Office Hysteroscopy for Reducing Pain and Anxiety
Brief Title: Use of Nitrous Oxide During Office Hysteroscopy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maaynei Hayesha Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Tamar Zur, P.I Dr Tamar Tzur. Senior gynecologist at Maaynei Hayesha, Maaynei Hayesha Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 0002-24mhmc
Record Dates: First submitted 2025-06-30; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Abnormal Uterine Bleeding; Postmenopausal Bleeding; Endometrial Polyps; Retained Products of Conception; Uterine Fibroids; Intrauterine Adhesions
Keywords: Inhaled nitrous oxide; Office hysteroscopy; Pain management; Visual analogue scale (VAS); Anxiety reduction; Gynecology
MeSH Terms: conditions — Metrorrhagia; Leiomyoma; Gynatresia; Agnosia

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial of inhaled nitrous oxide vs inhaled ambient air
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment- inhaled nitrous oxide (Active Comparator): Participants in the Nitrous Oxide group will inhale a fixed 50:50 mixture of nitrous oxide (N₂O) and oxygen (O₂), starting one minute prior to the procedure and continuing throughout its duration.
  The gas is administered via a self-administered demand-valve face mask connected to the Blendox system (Ambulanc®, Italy).
  Interventions: Procedure: Inhalation of Nitrous Oxide (N₂O) during Office Operative Hysteroscopy
- Inhaled ambient air control group (Placebo Comparator): Participants in the control group will inhale ambient air starting one minute prior to the procedure and will continue inhalation throughout its duration.
  The ambient air is administered via a self-administered demand-valve face mask connected to the Blendox system (Ambulanc®, Italy).
  Interventions: Procedure: inhalation of ambient air during office hysteroscopy

INTERVENTIONS:
Procedure: Inhalation of Nitrous Oxide (N₂O) during Office Operative Hysteroscopy — Inhaled nitrous oxide
  Arms: treatment- inhaled nitrous oxide
Procedure: inhalation of ambient air during office hysteroscopy — inhalation of ambient air
  Arms: Inhaled ambient air control group

SUMMARY:
The goal of this clinical trial is to assess the use of inhaled nitrous oxide during office hysteroscopy.

The main questions it aims to answer are:

* Does it reduce pain during the procedure?
* Does it increase the success rate?
* Does it improve patient satisfaction?
* Does it reduce anxiety?
* Which populations benefit more (e.g., parity, menopausal status, number of previous surgeries, type and duration of procedure, and type of device)?

Participants will be asked about their pain levels during the procedure, as well as their anxiety levels. All responses will be recorded.

Written informed consent will be obtained prior to initiation.

DETAILED DESCRIPTION:
Office hysteroscopy offers a convenient alternative to operating room-based procedures, yet many patients experience pain and anxiety significant enough to interfere with procedural completion. Nitrous oxide is a fast-acting inhaled agent with both analgesic and anxiolytic properties, widely used in outpatient settings across various medical specialties.

This study will investigate the role of nitrous oxide in improving patient tolerability and comfort during office hysteroscopy. Participants will undergo a standardized procedural protocol with either nitrous oxide or ambient air administered via a demand-valve mask system. Comprehensive data on patient responses during the procedure will be collected and analyzed.

The study will also examine variability in patient responses across different subgroups and procedural types. All procedures will adhere to ethical standards, and patient confidentiality will be maintained throughout.

ELIGIBILITY:
Inclusion Criteria:

Women aged ≥18 years Scheduled to undergo operative office hysteroscopy for clinical indications

Exclusion Criteria:

Any contraindications to N₂O, including:

Pneumothorax Significant chronic obstructive pulmonary disease (COPD) Upper airway obstruction Bowel obstruction Middle ear pathology (e.g., recent ear surgery or active ear infection) Severe recent intraocular gas injection Severe vitamin B12 deficiency Known hypersensitivity to N₂O

Women who will decline randomization or unable to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified females assigned female at birth are eligible to participate.
Enrollment: 400 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of Pain During Office Hysteroscopy Between Inhaled Nitrous Oxide (Treatment Group) and Ambient Air (Placebo Group) | Periprocedural (start to end of the hysteroscopy procedure)
  The difference in pain between the two groups will be assessed using the Visual Analog Scale (VAS), ranging from 0 to 10, where 0 indicates no pain and 10 represents the worst imaginable pain.
  Pain scores will be collected at three time points throughout the procedure
  : uterine entry, during the procedure, and immediately after its completion.

SECONDARY OUTCOMES:
Incidence of side effects related to inhaled substance | Periprocedural (start to end of the hysteroscopy procedure)
  The number and type of side effects reported during the procedure following administration of the inhaled agent (nitrous oxide or ambient air), including nausea, dizziness and presyncope. Adverse events will be recorded and categorized.
Procedure completion | Periprocedural
  Success is defined as the completion of the planned hysteroscopy procedure without the need for an additional intervention - either a repeat hysteroscopy or transfer to the operating room.
  The outcome will be measured as the percentage of participants for whom the procedure was successfully completed as planned.
Patient satisfaction with the procedure | Immediately post-procedure
  Assessed after the procedure by a binary question: "Would you be willing to undergo the same procedure again with the same inhaled agent?" (Yes/No)

OTHER OUTCOMES:
Subgroup differences in pain reduction associated with nitrous oxide during office hysteroscopy | Periprocedural (start to end of the hysteroscopy procedure)
  To evaluate whether specific patient characteristics are associated with greater pain reduction from nitrous oxide use during office hysteroscopy.
  Subgroups include nulliparity, prior surgeries, prolonged procedure duration, type of procedure, and type of hysteroscopic device. Pain will be measured using visual analogue scale (VAS) ranging from 0 to 10, where 0 indicates no pain and 10 represents the worst imaginable pain. Assessments will be performed at three points: uterine entry, during the procedure and immediately after.
Pre-procedural anxiety level assessed using modified State-Trait Anxiety Inventory (STAI) | Immediately before the procedure
  Anxiety levels will be assessed prior to the start of the hysteroscopy using a modified version of the State-Trait Anxiety Inventory (STAI) questionnaire. This tool evaluates both:
  State anxiety (temporary emotional state) Trait anxiety (long-term anxiety disposition) The state subscale includes 5 items, and the trait subscale includes 4 items.
  Each item is scored on a 5-point Likert scale (1 to 5), where:
  1 = lowest anxiety 5 = highest anxiety Total scores are calculated separately for state and trait components. Higher scores indicate greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Tzur, MD, Principal Investigator — Mayanei Hayeshua Medical Center
Locations (1):
- Mayanei HaYeshua Medical Center, Bnei Brak, Israel

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including pain scores, anxiety scores, demographic characteristics, and procedural outcomes, will be made publicly available through an open-access data repository (e.g., Zenodo) at the time of primary results publication.
  The data will be freely accessible for academic and research use, with no restrictions or approval required.
Supporting Information: Study Protocol
Time Frame: De-identified individual participant data (IPD) and supporting information will be made publicly available at the time of primary results publication in a peer-reviewed journal.
  The data will remain accessible indefinitely via an open-access online repository.
Access Criteria: The IPD and supporting documents will be accessible to all users via open access. No request or approval will be required.
  A direct link to the data repository (e.g., Figshare, Zenodo) will be provided in the publication.

REFERENCES:
- [Background] Likis FE, Andrews JC, Collins MR, Lewis RM, Seroogy JJ, Starr SA, Walden RR, McPheeters ML. Nitrous oxide for the management of labor pain: a systematic review. Anesth Analg. 2014 Jan;118(1):153-67. doi: 10.1213/ANE.0b013e3182a7f73c. PMID 24356165
- [Background] Buhre W, Disma N, Hendrickx J, DeHert S, Hollmann MW, Huhn R, Jakobsson J, Nagele P, Peyton P, Vutskits L. European Society of Anaesthesiology Task Force on Nitrous Oxide: a narrative review of its role in clinical practice. Br J Anaesth. 2019 May;122(5):587-604. doi: 10.1016/j.bja.2019.01.023. Epub 2019 Feb 22. PMID 30916011
- See also: Similar study principle evaluating inhaled nitrous oxide vs oral analgesia during office hysteroscopy — https://doi.org/10.1016/j.contraception.2016.09.006